# **GENERAL INFORMED CONSENT FORM**

Official Study Title:

Comparison of Scoring Systems in Predicting Morbidity and Mortality in Patients Undergoing Gastrointestinal Malignancy Surgery

ClinicalTrials.gov Identifier:

NCTXXXXXXX (Not yet assigned)

Document Date: 27 January 2021

## Purpose of the Study

You are invited to participate in a research study titled "Comparison of Scoring Systems in Predicting Morbidity and Mortality in Patients Undergoing Gastrointestinal Malignancy Surgery." The purpose of this study is to evaluate and compare various perioperative risk scoring systems in predicting postoperative complications, morbidity, and mortality in patients undergoing gastrointestinal malignancy surgery under general anesthesia. A total of 120 patients are planned to be included in this study.

## **Voluntary Participation**

Your participation in this study is voluntary. You may refuse to participate or withdraw at any time without providing a reason. Your decision will not affect your medical care or your relationship with your healthcare team.

## Study Procedures

If you agree to participate, your preoperative medical history and postoperative symptoms will be recorded. No additional procedures beyond routine clinical care will be performed.

### Risks and Discomforts

There are no anticipated risks or discomforts associated with participation in this observational study.

#### Potential Benefits

This study may not provide direct benefit to you. However, the knowledge gained may contribute to improving perioperative risk prediction in gastrointestinal malignancy surgery.

# Costs and Compensation

There will be no financial cost to you for participating in this study, and no payment will be made.

## Confidentiality

All personal data will remain confidential and will be used only for research purposes. Identifying information will not be disclosed.

## **Contact Information**

For further information, you may contact Dr. Mehmet Emre Geçici at +90 216 458 30 00 / 31822.

# Participant Statement

I have read and understood the information provided above. I voluntarily agree to participate in this clinical research study.

| Participant | |
|-----------------------|---------|
| Name and Surname: | |
| Signature: | Date: |
| Physician Obtaining ( | Consent |
| Name, Surname, Title | e: |
| Signature: | Date: |